CLINICAL TRIAL: NCT04529616
Title: Single Center Exploratory Study To Evaluate The Use Of The RxSight Light Adjustable Lens (LAL) And The Light Delivery Device (LDD) To Improve Visual Outcomes
Status: Completed | Type: Interventional
Sponsor: RxSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-036
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Aphakia; Cataract
Keywords: Light Adjustable Lens; Intraocular lens; LAL
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Light adjustable lens (LAL) and Light Delivery Device (LDD) (Experimental)
  Interventions: Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD)

INTERVENTIONS:
Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD) — Eligible eyes will receive Light adjustable lens with Light delivery Device treatments

SUMMARY:
The objective of this study is to evaluate, for the visual correction of aphakia, whether the RxSight Light Adjustable Lens (LAL) and Light Delivery Device (LDD) can be used to improve visual outcomes after performing adjustments of the LAL with the LDD. This is an exploratory study. No primary effectiveness endpoints will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Must sign a written Informed Consent form and be willing to undergo cataract surgery for unilateral or bilateral implantation of the RxLAL.
* Age 30 or older on the day the cataract surgery is performed.
* Study eye must have cataract causing reduction in best corrected distance visual acuity (BCDVA) to a level of 20/32 or worse with or without a glare source.
* Willing and able to comply with the requirements for study specific procedures and visits.

Exclusion Criteria:

* Study eye with zonular laxity or dehiscence.
* Study eye with diabetes with any evidence of retinopathy.
* Study eye with history of uveitis.
* Subjects taking systemic medication that may increase sensitivity to UV light such as tetracycline, doxycycline, psoralens, amiodarone, phenothiazines, chloroquine, hydrochlorothiazide, hypericin, ketoprofen, piroxicam, lomefloxacin, and methoxsalen. LDD treatment in patients taking such medications may lead to irreversible phototoxic damage to the eye. This is only a partial list of photosensitizing medications. Please evaluate all medications that the patient is taking for this effect prior to consideration for implantation.
* Subjects taking a systemic medication that is considered toxic to the retina such as tamoxifen.
* Study eye with history of ocular herpes simplex virus.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CODET Vision Institute, Tijuana, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
Started | 79; 141 Eyes
Completed | 79; 141 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 59
  Black | 0
  Other | 0
  Not Reported | 20
Region of Enrollment [Number; unit: participants]
  Mexico | 79

OUTCOME MEASURES:

1. Primary Outcome: Percent of Eyes With Uncorrected Distance Visual Acuity (UCDVA) of 20/20 or Better
Description: Values were measured via Early Treatment Diabetic Retinopathy Study (ETDRS) testing.
Time Frame: 3 months post op
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
Number analyzed (Participants) | 32
Number analyzed (Eyes) | 32
Eyes | 21

2. Primary Outcome: Proportion of Eyes Simultaneously With (1) Monocular UCDVA of 20/25 or Better and (2) Monocular Uncorrected Intermediate Visual Acuity (UCIVA) of 20/32 or Better and (3) Monocular Uncorrected Near Visual Acuity (UCNVA) of 20/40 or Better
Description: Visual performance parameters will be collected and summarized for eyes that received a presbyopia adjustment
Time Frame: 12 months post op
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
Number analyzed (Participants) | 79
Number analyzed (Eyes) | 95
Eyes | 91

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
All-Cause Mortality (participants affected / at risk) | 1/79
Serious Adverse Events (participants affected / at risk) | 2/79
Other Adverse Events (participants affected / at risk) | 9/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) (N=79)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Blood clots secondary to head trauma from a fall (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) (N=79)
Intraretinal microhemorrhage secondary to diabetes and hypertension (Eye disorders) | 1 (1)
Microaneurism, intraretinal hemorrhage dots secondary to history of diabetes (Eye disorders) | 1 (1)
Corneal epithelium: epithelialized with SPK (Eye disorders) | 1 (2)
Granular deposits over IOL (Eye disorders) | 1 (2)
Epiretinal membrane (Eye disorders) | 3 (4)
Drusen (Eye disorders) | 2 (4)
Pigmentary changes (Eye disorders) | 1 (1)
Optic nerve edema secondary to head trauma (Nervous system disorders) | 1 (1)
Posterior capsular opacity (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT04529616/Prot_SAP_000.pdf